CLINICAL TRIAL: NCT03070470
Title: Comprehensive in Vitro Proarrhythmia Assay (CiPA) Clinical Phase 1 ECG Biomarker Validation Study (CiPA Phase 1 ECG Biomarker Study)
Brief Title: CiPA Phase 1 ECG Biomarker Validation Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 16-086D; SCR-004 (Other: Spaulding Clinical Research LLC)
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Drug-induced QT Prolongation; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Ranolazine; Verapamil; Lopinavir; Chloroquine; dofetilide; Diltiazem

STUDY DESIGN:
Intervention Model Description: This clinical study consists of 2 parts:
  * 50 subjects in Part 1 will be randomized to receive one of four drugs (ranolazine, verapamil, lopinavir / ritonavir, chloroquine) or placebo over 3 days.
  * 10 subjects in Part 2 will be randomized to receive one of two treatment sequences (1. dofetilide or 2. diltiazem combined with dofetilide) over 3 days, then after washout, the subjects will receive the other treatment sequence over 3 days. Thus, Part 2 will have a cross-over component.
  A maximum of 14 additional replacement subjects may be enrolled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Ranolazine (Active Comparator): Ranolazine 1500 mg two times per day for 2.5 days
  Interventions: Drug: Ranolazine
- Verapamil (Active Comparator): Verapamil 120 mg immediate release (IR) morning and afternoon doses on Days 1 and 2, 240 mg extended release (ER) evening dose on Days 1 and 2, and 120 mg IR morning dose on Day 3
  Interventions: Drug: Verapamil
- Lopinavir / Ritonavir (Active Comparator): Lopinavir / Ritonavir 800 mg / 200 mg two times per day for 2.5 days
  Interventions: Drug: Lopinavir / Ritonavir
- Chloroquine (Active Comparator): Chloroquine 1000 mg on Day 1, 500 mg on Day 2, 1000 mg on Day 3
  Interventions: Drug: Chloroquine
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo
- Dofetilide and Diltiazem (Active Comparator): In one period subjects receive Dofetilide 0.125 mg on Day 1, 0.375 mg on Day 3.
  In a second period (randomized cross-over) subject receive Diltiazem 120 mg IR morning dose on Day 8, 240 mg ER evening dose on Days 8 and 9, and 120 mg IR on Day 10 with coadministration of 0.25 mg dofetilide on Day 10.
  Interventions: Drug: Dofetilide and Diltiazem

INTERVENTIONS:
Drug: Ranolazine — Ranolazine 1500 mg orally two times per day for 2.5 days
  Arms: Ranolazine
Drug: Verapamil — Verapamil 120 mg immediate release (IR) morning and afternoon doses on Days 1 and 2, 240 mg extended release (ER) evening dose on Days 1 and 2, and 120 mg IR morning dose on Day 3 (all oral doses)
  Arms: Verapamil
Drug: Lopinavir / Ritonavir — Lopinavir / Ritonavir 800 mg / 200 mg orally two times per day for 2.5 days
  Arms: Lopinavir / Ritonavir
Drug: Chloroquine — Chloroquine 1000 mg on Day 1, 500 mg on Day 2, 1000 mg on Day 3 (all oral doses)
  Arms: Chloroquine
Drug: Placebo — Placebo (administered orally)
  Arms: Placebo
Drug: Dofetilide and Diltiazem — In one period subjects receive Dofetilide 0.125 mg on Day 1, 0.375 mg on Day 3.
  In a second period (randomized cross-over) subject receive Diltiazem 120 mg IR morning dose on Day 8, 240 mg ER evening dose on Days 8 and 9, and 120 mg IR on Day 10 with coadministration of 0.25 mg dofetilide on Day 10.
  Arms: Dofetilide and Diltiazem

SUMMARY:
This study will assess whether exposure response analysis of the electrocardiographic QTc and J-Tpeakc intervals in Phase 1 clinical pharmacology studies can be used to confirm that drugs that predominantly block the potassium channel encoded by the human ether-à-go-go-related gene (hERG) with approximately equipotent late sodium and/or calcium block ("balanced ion channel" drugs) do not cause J-Tpeakc prolongation and that drugs that predominantly block hERG without late sodium or L-type calcium current block ("predominant hERG" drugs) cause QTc prolongation.

DETAILED DESCRIPTION:
This study will assess whether exposure response analysis of the electrocardiographic QTc and J-Tpeakc intervals in Phase 1 clinical pharmacology studies can be used to confirm that "balanced ion channel" drugs do not cause J-Tpeakc prolongation and that "predominant hERG" drugs cause QTc prolongation. This clinical study consists of 2 parts: a 50-subject parallel part (Part 1) and a 10-subject crossover part (Part 2). Up to 74 healthy subjects will be enrolled (including 14 potential replacement subjects).

Part 1 will be a double-blind, randomized, placebo-controlled, 1 period parallel design to assess the effect of 4 marketed drugs and 1 placebo on the QTc and J-Tpeakc intervals in 50 healthy subjects. A parallel design similar to a single or multiple ascending dose (SAD/MAD) Phase 1 study will be used that will result in each study drug being administered to 10 subjects, and placebo to 10 subjects, in 1 period of 3 consecutive days to achieve low and high drug exposure.

Part 2 will be a double-blind, randomized, 2-period crossover design to assess the effect of hERG block (dofetilide) versus calcium block (diltiazem) on the QTc and J-Tpeakc intervals in 10 healthy subjects on Days 1, 2, and 3 (Period 1) and Days 8, 9, and 10 (Period 2).

ELIGIBILITY:
Inclusion criteria:

1. Subject signs an institutional review board (IRB) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act [HIPAA] authorization) before any study related procedures are performed.
2. Subject is a healthy man or woman, 18 to 50 years of age, inclusive, who weighs at least 50 kg (110 pounds) and has a body mass index of 18 to 30 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead ECG results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Female subjects will be at least 2 years postmenopausal, surgically sterile, or practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique).
5. Female subjects must not be pregnant or lactating before enrollment in the study.
6. Male or female subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from Screening until 30 days after the last dose of study drug.
7. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion criteria:

1. Subject has a safety 12 lead ECG result at Screening or Check in with evidence of any of the following abnormalities:

   * QTc using Fridericia correction (QTcF) >430 msec
   * PR interval >220 msec or <120 msec
   * QRS duration >110 msec
   * Second- or third-degree atrioventricular block
   * Complete left or right bundle branch block or incomplete right bundle branch block
   * Heart rate <50 or >90 beats per minute
   * Pathological Q-waves (defined as Q wave >40 msec)
   * Ventricular pre-excitation
2. Subject has more than 12 ectopic beats during the 3 hour Holter ECG at Screening.
3. Subject has a history of unexplained syncope, structural heart disease, long QT syndrome, heart failure, myocardial infarction, angina, unexplained cardiac arrhythmia, torsade de pointes, ventricular tachycardia, or placement of a pacemaker or implantable defibrillator. Subjects will also be excluded if there is a family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative due to cardiac causes at a young age) or Brugada syndrome.
4. Subject has a history or current evidence of any clinically significant (as determined by the investigator) cardiovascular, dermatologic, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, neurologic, psychiatric, pulmonary, renal, urologic, and/or other major disease or malignancy (excluding nonmelanoma skin cancer). The investigator may allow exceptions to these criteria (e.g., cholecystectomy, childhood asthma) following discussion with the medical monitor.
5. Subject has a history of thoracic surgery.
6. Subject has any condition possibly affecting study drug absorption (e.g., gastrectomy, Crohn's disease, irritable bowel syndrome).
7. Subject has a skin condition likely to compromise ECG electrode placement.
8. Subject is a female with breast implants.
9. Subject's laboratory test results at Screening or Check in are outside the reference ranges provided by the clinical laboratory and considered clinically significant (as determined and documented by the investigator or designee).
10. Subject's laboratory test results at Screening or Check in indicate hypokalemia, hypocalcemia, or hypomagnesemia according to lower limits of the reference ranges provided by the clinical laboratory.
11. Subject's laboratory test results at Screening or Check in are >2 × the upper limit of normal (ULN) for alanine aminotransferase or aspartate aminotransferase, >1.5 × ULN for bilirubin, or >1.5 × ULN for creatinine.
12. Subject has a positive test result at Screening for human immunodeficiency virus I or II antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
13. Subject has a mean systolic blood pressure <100 or >140 mmHg or a mean diastolic blood pressure <50 or >90 mmHg at either Screening or Check in. Blood pressure will be measured in triplicate after the subject has been resting in a supine position for a minimum of 5 minutes.
14. Subject has a known hypersensitivity to any of the study drugs or related compounds.
15. Subject has consumed alcohol, xanthine containing products (e.g., tea, coffee, chocolate, cola), caffeine, grapefruit, or grapefruit juice within 48 hours before dosing or anticipates an inability to abstain from these products throughout the duration of the study.
16. Subject has used nicotine containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks before Screening (self reported).
17. Subject is unable to tolerate a controlled, quiet, study conduct environment, including avoidance of music, television, movies, games, and activities that may cause excitement, emotional tension, or arousal during the prespecified time points (e.g., before and during ECG extraction windows).
18. Subject is unwilling to comply with study rules, including the study-specific diet, attempting to void at specified times (e.g., before ECG extraction windows), remaining quiet, awake, undistracted, motionless, and supine during specified times, and avoiding vigorous exercise as directed.
19. Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months before Screening, has a history of alcoholism or drug/chemical/substance abuse within 2 years before Screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine, or 1 ounce of spirits/hard liquor), or has a positive test result for alcohol or drugs of abuse at Screening or Check in.
20. Subject has used any prescription or nonprescription drugs (including aspirin or nonsteroidal anti inflammatory drugs [NSAIDs] and excluding oral contraceptives and acetaminophen) within 14 days or 5 half lives (whichever is longer), or complementary and alternative medicines within 28 days before the first dose of study drug.
21. Subject is currently participating in another clinical study of an investigational drug or has been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of the compound.
22. Subject has had any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days before Check in.
23. Subject has any other condition that precludes his or her participation in the study (as determined by the investigator).
24. Subject is unwilling to have genetic analysis performed or a blood sample collected for isolating peripheral blood mononuclear cells (PBMCs).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan released as supplementary materials together with study design and rationale manuscript. ECG analysis plan published together with an update of the CiPA initiative. Annotated ECG waveforms, pharmacokinetic, and other subject level clinical data released as ECGCIPA database in PhysioNet. Clinical study report and analytic code released as supporting information (i.e., study results report) of study results manuscript. See references section.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: January 2018: Study protocol and SAP (doi: 10.1002/cpt.896).
  August 2018: ECG analysis plan (doi: 10.1016/j.jelectrocard.2018.08.003).
  December 2018: Annotated ECG waveforms and clinical data database (https://physionet.org/physiobank/database/ecgcipa/)
  December 2018: Study results report published (doi: 10.1002/cpt.1303)
Access Criteria: Open access
URL: https://physionet.org/physiobank/database/ecgcipa/

REFERENCES:
- [Background] Vicente J, Zusterzeel R, Johannesen L, Mason J, Sager P, Patel V, Matta MK, Li Z, Liu J, Garnett C, Stockbridge N, Zineh I, Strauss DG. Mechanistic Model-Informed Proarrhythmic Risk Assessment of Drugs: Review of the "CiPA" Initiative and Design of a Prospective Clinical Validation Study. Clin Pharmacol Ther. 2018 Jan;103(1):54-66. doi: 10.1002/cpt.896. Epub 2017 Nov 16. PMID 28986934
- [Background] Vicente J. Update on the ECG component of the CiPA initiative. J Electrocardiol. 2018 Nov-Dec;51(6S):S98-S102. doi: 10.1016/j.jelectrocard.2018.08.003. Epub 2018 Aug 7. PMID 30121123
- [Result] Vicente J, Zusterzeel R, Johannesen L, Ochoa-Jimenez R, Mason JW, Sanabria C, Kemp S, Sager PT, Patel V, Matta MK, Liu J, Florian J, Garnett C, Stockbridge N, Strauss DG. Assessment of Multi-Ion Channel Block in a Phase I Randomized Study Design: Results of the CiPA Phase I ECG Biomarker Validation Study. Clin Pharmacol Ther. 2019 Apr;105(4):943-953. doi: 10.1002/cpt.1303. Epub 2019 Jan 18. PMID 30447156
- Available data/document: Individual Participant Data Set: ECGCIPA — https://physionet.org/physiobank/database/ecgcipa/ — ECG effects of ranolazine, verapamil, lopinavir+ritonavir, chloroquine, dofetilide, diltiazem, and dofetilide+diltiazem in a small sample size clinical study. The ECGCIPA database contains multi-channel ECG recordings, pharmacokinetic, and clinical data of 60 subjects participating in the CiPA ECG validation study.

RESULTS

PARTICIPANT FLOW:
Groups:
- Dofetilide and Diltiazem: In one period subjects receive Dofetilide 0.125 mg on Day 1, 0.375 mg on Day 3.
  In a second period (randomized cross-over) subject receive Diltiazem 120 mg IR morning dose on Day 8, 240 mg ER evening dose on Days 8 and 9, and 120 mg IR on Day 10 with coadministration of 0.25 mg dofetilide on Day 10.
  Dofetilide and Diltiazem: In one period subjects receive Dofetilide 0.125 mg on Day 1, 0.375 mg on Day 3.
  In a second period (randomized cross-over) subject receive Diltiazem 120 mg IR morning dose on Day 8, 240 mg ER evening dose on Days 8 and 9, and 120 mg IR on Day 10 with coadministration of 0.25 mg dofetilide on Day 10.
Period: Overall Study
Arm/Group | Ranolazine | Verapamil | Lopinavir / Ritonavir | Chloroquine | Placebo | Dofetilide and Diltiazem
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 9 | 10 | 10 | 10 | 8
Not Completed | 0 | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Verapamil | Lopinavir / Ritonavir | Chloroquine | Placebo | Dofetilide and Diltiazem | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (8.0) | 28.2 (7.9) | 32.6 (11.1) | 28.8 (8.8) | 33.3 (9.0) | 33.4 (7.2) | 31.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6 | 3 | 2 | 5 | 22
  Male | 8 | 6 | 4 | 7 | 8 | 5 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 10 | 9 | 10 | 9 | 8 | 9 | 55
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 5 | 7 | 5 | 4 | 32
  White | 3 | 4 | 5 | 2 | 4 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 10 | 10 | 10 | 10 | 60
Weight [Mean (Standard Deviation); unit: Kg] | 80.3 (11.1) | 77.1 (10.2) | 76.2 (6.1) | 72.4 (11.3) | 77.5 (15.6) | 69.5 (9.4) | 75.5 (11.1)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 116.6 (9.5) | 109.2 (6.6) | 119.4 (10.0) | 114.8 (8.1) | 116.6 (6.4) | 113.4 (8.2) | 115.0 (8.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 66.7 (8.7) | 63.4 (6.9) | 67.3 (8.5) | 66.9 (5.5) | 66.7 (9.0) | 64.2 (6.9) | 65.9 (7.5)
Heart Rate [Mean (Standard Deviation); unit: BPM] | 59.8 (8.9) | 63.6 (9.8) | 61.3 (9.3) | 59.2 (9.5) | 58.6 (5.6) | 61.9 (6.1) | 60.7 (8.2)
PR Interval [Mean (Standard Deviation); unit: ms] | 182.4 (23.9) | 178.4 (16.2) | 162.3 (16.5) | 159.1 (15.5) | 164.4 (15.0) | 171.6 (19.4) | 169.7 (19.2)
QRS Duration [Mean (Standard Deviation); unit: ms] | 90.1 (7.7) | 82.9 (8.2) | 87.1 (5.8) | 84.7 (6.7) | 85.4 (11.5) | 87.3 (9.4) | 86.3 (8.4)
QTc (Fridericia's heart rate corrected QT interval) [Mean (Standard Deviation); unit: ms] | 386.0 (20.2) | 386.5 (17.8) | 383.9 (17.1) | 393.3 (20.0) | 387.1 (13.7) | 397.1 (26.1) | 389.0 (19.2)
J-Tpeakc (heart rate corrected J-Tpeak interval) [Mean (Standard Deviation); unit: ms] | 227.7 (22.7) | 239.4 (22.4) | 231.0 (14.5) | 238.7 (20.3) | 229.5 (24.2) | 239.7 (29.4) | 234.3 (22.3)
Tpeak-Tend interval [Mean (Standard Deviation); unit: ms] | 68.7 (7.9) | 65.1 (6.6) | 65.7 (7.9) | 69.7 (8.7) | 72.5 (6.4) | 70.6 (14.8) | 68.7 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline J-Tpeakc With "Balanced Ion Channel" Drugs (Ranolazine, Verapamil, Lopinavir / Ritonavir)
Description: The primary outcome measure for the "balanced ion channel" drugs (ranolazine, verapamil, lopinavir / ritonavir) is for the upper bound of the 2-sided 90% confidence interval (CI) to be <10 msec for the projected placebo-corrected change from baseline J-Tpeakc effect at the peak plasma level on Day 3 using a linear mixed-effects exposure response model. Placebo drug concentration was set to 0 (see SAP).
Time Frame: 3 days
Population: Placebo data was used in the statistical analysis to account for placebo effect. Chloroquine, and dofetilide and diltiazem data were collected but not part of the primary J-Tpeakc analysis. The underlying raw data (available at https://doi.org/10.13026/C2967M) were the input in the statistical analysis. Summary included per PRS review team request.
Measure: Median (Full Range); unit: ms
Arm/Group | Ranolazine | Verapamil | Lopinavir / Ritonavir | Chloroquine | Placebo | Dofetilide and Diltiazem
Number analyzed (Participants) | 10 | 10 | 10 | 0 | 10 | 0
ms | -8.3 [-66.4 to 23.6] | -7.8 [-58.1 to 11.4] | -11.5 [-50.7 to 47.4] |  | -10.9 [-81.2 to 14.7] |
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Upper bound of the 2-sided 90% confidence interval (CI) to be <10 msec for the projected placebo-corrected change from baseline J-Tpeakc effect at the peak plasma level on Day 3 using a linear mixed-effects exposure response model; Test type: Other — The appropriateness of the linear model will be assessed. Projected estimates will be computed only if the linear model is found acceptable; Mixed Models Analysis — The degrees of freedom for the model estimates were determined by the Kenward-Rogers method as prespecified in the SAP; Mean Difference (Final Values) = 1.2, 90% CI 2-sided [-9.5 to 12.0]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; The degrees of freedom for the model estimates were determined by the Kenward-Rogers method as prespecified in the SAP; Mean Difference (Final Values) = -2.6, 90% CI 2-sided [-11.4 to 6.1]
Statistical Analysis 3: Comparison: Lopinavir / Ritonavir vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; The degrees of freedom for the model estimates were determined by the Kenward-Rogers method as prespecified in the SAP; Mean Difference (Final Values) = -2.9, 90% CI 2-sided [-14.6 to 8.8]

2. Primary Outcome: Change From Baseline QTc With "Predominant hERG" Blocking Drug (Chloroquine)
Description: The primary outcome measure for the "predominant hERG" drug (chloroquine) is for the upper bound of the 2-sided 90% CI to be ≥10 msec for the projected placebo-corrected change from baseline QTc effect at the peak plasma level on Day 1 using a linear mixed-effects exposure response model
Time Frame: 3 days
Population: Ranolazine, verapamil, lopinavir/ritonavir, and dofetilide and diltiazem data were collected but not part of the primary QTc analysis. The underlying raw data (available at https://doi.org/10.13026/C2967M) were the input in the statistical analysis. Median and range summary included per PRS review team request.
Measure: Median (Full Range); unit: ms
Arm/Group | Ranolazine | Verapamil | Lopinavir / Ritonavir | Chloroquine | Placebo | Dofetilide and Diltiazem
Number analyzed (Participants) | 0 | 0 | 0 | 10 | 10 | 0
ms |  |  |  | 17.7 [-24.3 to 71.9] | -9.3 [-48.3 to 27.6] |
Statistical Analysis 1: Comparison: Chloroquine vs Placebo; Upper bound of the 2-sided 90% CI to be ≥10 msec for the projected placebo-corrected change from baseline QTc effect at the peak plasma level on Day 1 using a linear mixed-effects exposure response model; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; The degrees of freedom for the model estimates were determined by the Kenward-Rogers method as prespecified in the SAP; Mean Difference (Final Values) = 30.7, 90% CI 2-sided [22.6 to 38.9]

3. Primary Outcome: QTc Shortening From Calcium Block (Diltiazem) in the Presence of hERG Block (Dofetilide)
Description: * It will be assessed whether the projected QTc effect of dofetilide alone is significantly greater (i.e., p<0.05) than the projected QTc effect of the combination of dofetilide + diltiazem. This will be assessed at the dofetilide peak plasma level on Day 3 (computed from the combination of dofetilide + diltiazem) on the pooled dofetilide alone, diltiazem alone, and dofetilide + diltiazem data using a linear mixed effects model.
  * Subsequently, and if the test is significant for QTc, the same test will be performed to assess calcium block (diltiazem) effects on J-Tpeakc.
Time Frame: 3 days
Population: QTc, J-Tpeakc, and drug concentration data from all subjects in the dofetilide and diltiazem arm. Ranolazine, verapamil, lopinavir/ritonavir, chloroquine, and placebo data were collected but not part of this analysis (see SAP). The underlying raw data were the input in the statistical analysis. Summary included per PRS review team request.
Measure: Median (Full Range); unit: ms
Groups:
- Dofetilide: Data from the Dofetilide alone period of the crossover part:
  In one period subjects receive Dofetilide 0.125 mg on Day 1, 0.375 mg on Day 3.
  In a second period (randomized cross-over) subject receive Diltiazem 120 mg IR morning dose on Day 8, 240 mg ER evening dose on Days 8 and 9, and 120 mg IR on Day 10 with coadministration of 0.25 mg dofetilide on Day 10.
- Diltiazem+Dofetilide: Data from the diltiazem and dofetilide period of the crossover part:
  In one period subjects receive Dofetilide 0.125 mg on Day 1, 0.375 mg on Day 3.
  In a second period (randomized cross-over) subject receive Diltiazem 120 mg IR morning dose on Day 8, 240 mg ER evening dose on Days 8 and 9, and 120 mg IR on Day 10 with coadministration of 0.25 mg dofetilide on Day 10.
Arm/Group | Ranolazine | Verapamil | Lopinavir / Ritonavir | Chloroquine | Placebo | Dofetilide | Diltiazem+Dofetilide
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 10
ms |  |  |  |  |  | 2.2 [-35.2 to 64.5] | -1.7 [-31.9 to 53.6]

ADVERSE EVENTS:
Time Frame: 4 days
Description: MedDRA
Arm/Group | Ranolazine | Verapamil | Lopinavir / Ritonavir | Chloroquine | Placebo | Dofetilide and Diltiazem
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 5/10 | 9/10 | 4/10 | 2/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=10) | Verapamil (N=10) | Lopinavir / Ritonavir (N=10) | Chloroquine (N=10) | Placebo (N=10) | Dofetilide and Diltiazem (N=10)
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0
Abdominal Distention (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cold Sweat (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Decreased Appetite (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 5 | 1 | 1 | 0
Dissociation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dry Mouth (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Headache (General disorders) | 0 | 2 | 5 | 1 | 0 | 3
Menstrual Discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Nausea (General disorders) | 0 | 0 | 4 | 1 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Presyncope (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Somnolence (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vessel Puncture Site Pain (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 1
Vessel Puncture Site Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vessel Puncture Site Swelling (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT03070470/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03070470/SAP_001.pdf